CLINICAL TRIAL: NCT03926962
Title: Double-Blind, Randomized, Placebo-Controlled Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of Single Ascending Doses And The Effect Of Food On Oral WCK 4873 In Healthy Adult Volunteers
Brief Title: The Safety, Tolerability And Pharmacokinetics Of Single Ascending Doses And The Effect Of Food On Oral WCK 4873 In Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: W 4873 01
Record Dates: First submitted 2019-04-03; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — nafithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- WCK 4873 (Experimental): 100 to 1200 mg in tablets (the 100 mg dose cohort will receive half a tablet; higher dose cohorts will receive 1 or more tablets)
  Interventions: Drug: WCK 4873
- Placebo (Placebo Comparator): Visually matching placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: WCK 4873 — 100 to 1200 mg in tablets (the 100 mg dose cohort will receive half a tablet; higher dose cohorts will receive 1 or more tablets)
  Arms: WCK 4873
Drug: Placebo Oral Tablet — Visually matching placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled study, consisting of a single ascending dose (SAD) part and a 2-way crossover food effect (FE) part. Each subject will participate in only one cohort during the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI : 18-30 kg/m2 (Body Mass Index [BMI] [kg/m2] = Body weight [kg] Height2 [m2])
* Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "powerdrinks"), grapefruit (juice) from 48 h prior to entry in the clinical research center until discharge
* Medical history without major pathology

Exclusion Criteria:

* Evidence of clinically relevant pathology
* Mental handicap
* History of relevant drug and/or food allergies
* Regular/routine treatment with non-topical medications within 30 days prior to entry into the clinical research center
* Smoking within 60 days prior to drug administration and through the follow-up visit
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2013-06-25 (Actual); Study Completion 2013-07-13 (Actual)

PRIMARY OUTCOMES:
Assessing incidence of treatment emergent AEs | Day 18
  Incidence of treatment emergent AEs, abnormal clinical laboratory findings, variations in LFTs, abnormal physical examination findings, variations in vital signs and variations in 12-lead ECG
Evaluating PK parameters for profiling | Day 4
  plasma PK parameters -Area under curve (AUC0-t, AUC0-12, AUC0-24, AUC0-inf, %AUC)
Evaluating PK parameters for profiling | Day 4
  plasma PK parameters- maximum concentration (Cmax, Clast)
Evaluating PK parameters for profiling | Day 4
  plasma PK parameters tmax, tlast, kel, t½,
Evaluating PK parameters for profiling | Day 4
  urine PK paramters (Aeurine)
Evaluating PK parameters for profiling | Day 4
  feces PK paramters ( Aefeces)
Evaluating PK parameters for profiling | Day 4
  PMN white blood cell concentrations of WCK 4873.